CLINICAL TRIAL: NCT03462784
Title: Prevalance and Risk Factors for Complications in Children With B- Thalassemia Major
Brief Title: Complications in Children With B- Thalassemia Major
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tahany Naeem Saied Matta, Principal Investigator, Assiut University
Other Study IDs: Prev TM
Record Dates: First submitted 2018-02-23; First posted 2018-03-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Beta-thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — Demography; Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases
  Interventions: Other: Demographic, physical examination, data will becollected .

INTERVENTIONS:
Other: Demographic, physical examination, data will becollected . — Demographic data collected includ clinical diagnosis, sex, race, genotype, and phenotype.
  Historical data included information regarding immunizations, infection exposures, surgical procedures, organ dysfunction(Organ dysfunction was defined as a history of requiring medical treatment for heart disease, diabetes (Type 1 or 2), hypoparathyroidism, hypothyroidism, growth hormone deficiency, or gonadal failure) age at transfusion initiation, chelation therapy, type of RBC product, transfusion reactions, and antigen matching. Data will be collected from chart review, patient interviews, blood banking records, and laboratory

SUMMARY:
Worldwide, there are more than 60,000 births annually of serious forms of thalassemia .The World Health Organization considers thalassemia to be a major health burden.

Beta- thalassemia is a group of recessively inherited disorders of hemoglobin synthesis characterized by reduced synthesis of the ß-globin chain caused by a mutation. The homozygous state results in severe anemia which needs regular blood transfusion.

DETAILED DESCRIPTION:
Thalassemia is the most common monogenic disorder in the world .Thalassemia major (beta-thalassemia) affects a significant segment of the population in certain areas of the world. Alterations in migration patterns have changed the geographic distribution of this disease and made it a worldwide health problem with a high frequency in Africa, India, Southeast Asia and the Mediterranean area.

The combination of transfusion and chelation therapy has dramatically extended the life expectancy of these patients, thus transforming thalassemia from a rapidly fatal disease of childhood to a chronic illness compatible with a prolonged life. On the other hand, frequent blood transfusions leading to iron overload and the chronic nature of the disease have contributed to a whole new spectrum of complications in adolescents and young adults suffering from thalassemia major.

Complications associated with beta thalassemia, aside from the aforementioned anemia, are as follows

* Extramedullary hematopoiesis
* Asplenia secondary to splenectomy
* Medical complications from long-term transfusional therapy - Iron overload and transfusion-associated infections (eg, hepatitis) Increased risk for infections resulting from asplenia (eg, encapsulated organisms such as pneumococcus) or from iron overload (eg, Yersinia species))
* Cholelithiasis (eg, bilirubin stones) Study of the prevelance and risk fators responsible for thalassemia complication can help in adopting appropriating strategies for management of these complication.

ELIGIBILITY:
Inclusion Criteria

* All patient from 1 year up to 18 year (1year-18 year) admitted at Haematology unit at Assuit University Children Hospital who were diagnosed as Beta thalassemia major

Exclusion Criteria:

* Age less than 1 year( 1 ≤ year)
* Children who diagnosed as other types of thalassemia except Beta thalassemia major

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who diagnosed as B thalassemia major
Sampling Method: Non-Probability Sample
Enrollment: 201 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevelance of Comlications of Beta -Thalassemia major in children | one year
  Demographic data collected includ clinical diagnosis, sex, race, genotype, and phenotype.
  Historical data included information regarding immunizations, infection exposures, surgical procedures, organ dysfunction (Organ dysfunction was defined as a history of requiring medical treatment for heart disease, diabetes (Type 1 or 2), hypoparathyroidism, hypothyroidism, growth hormone deficiency, or gonadal failure) age at transfusion initiation, chelation therapy, type of RBC product, transfusion reactions, and antigen matching. Data will be collected from chart review, patient interviews, blood banking records, and laboratory testing. All these data will be collected to know the type of complication and measure the prevelance of these complication

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Modell B, Darlison M. Global epidemiology of haemoglobin disorders and derived service indicators. Bull World Health Organ. 2008 Jun;86(6):480-7. doi: 10.2471/blt.06.036673. PMID 18568278
- [Result] Weatherall DJ. The inherited diseases of hemoglobin are an emerging global health burden. Blood. 2010 Jun 3;115(22):4331-6. doi: 10.1182/blood-2010-01-251348. Epub 2010 Mar 16. PMID 20233970